CLINICAL TRIAL: NCT03918122
Title: Master Preceptor Fellowship Program: A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Not enough enrolled
Sponsor: Pacific Northwest University of Health Sciences (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, PNWU OSA, Principal Investigator, Pacific Northwest University of Health Sciences
Other Study IDs: 2018-025
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Self-Assessment; Knowledge, Attitudes, Practice
Keywords: Preceptor; Physician Leadership; Medical Education
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-Assessment via pre and post survey — Master Preceptor Fellows will assess and evaluation professional development, knowledge, clinical practices and master preceptor knowledge before the Master Preceptor Fellowship and After completion of the Master Preceptor Fellowship

SUMMARY:
The Master Preceptor Fellowship Pilot Study is a prospective cohort study that is being conducted to measure changes in participant knowledge, teaching efficacy, leadership skills, job satisfaction and quality of life.

DETAILED DESCRIPTION:
The Master Preceptor Fellows are physicians or physician assistants who have worked in primary care setting for a minimum of one year. The participants agree to participate in a 52-week (1-year) program designed to enhance the primary care physician's knowledge and skills via self-directed and didactic coursework along with a transformational community-based project. The culmination of the mentorship, leadership, and educational experiences gained in the Master Preceptor Fellowship (MPF) will allow the primary care physician champion to apply his or her innovative response to an identified need in their community.

ELIGIBILITY:
Inclusion Criteria:

* Have a medicine or physician assistant degree (MD/DO or PA)
* Be board certified or board eligible in family medicine, general internal medicine, or general -pediatrics; or be certified as a physician assistant
* Have a position in a community-based primary care site
* Have a record of practice in a primary care discipline field for at least two years
* Be at least 18 years of age

Exclusion Criteria:

* Unable to adequately speak and comprehend English
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians (MD or DO) or Physician Assistants (PA) that have been in practice for at least one year. Physicians must be board certified or board eligible in family medicine, general internal medicine or general pediatrics. Physician assistants must be certified as a physician assistant.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in Knowledge of Physician Teaching Self Efficacy (PTSQ) | Baseline to fellowship completion [approximately 52 weeks]
  The PTSQ survey measures a physician's belief to provide high quality clinical teaching when facing regularly occurring critical teaching situations. This is a 16 item survey with a rating scale of 0=Not applicable, 1=Somewhat does not apply, 2=Neutral, 3=Somewhat applies, 4=Applies completely. A higher score indicating a higher belief in one's ability to provide high quality clinical teaching in critical teaching situations.
Changes in Knowledge Physician Teaching Self Efficacy (PTSQ) | Fellowship completion [approximately 52 weeks] to 6 months post completion [approximately 77 weeks]
  The PTSQ survey measures a physician's belief to provide high quality clinical teaching when facing regularly occurring critical teaching situations. This is a 16 item survey with a rating scale of 0=Not applicable, 1=Somewhat does not apply, 2=Neutral, 3=Somewhat applies, 4=Applies completely. A higher score indicating a higher belief in one's ability to provide high quality clinical teaching in critical teaching situations.
Changes in Quality of Life (PROMIS Global Health Survey) | Baseline to fellowship completion [approximately 52 weeks]
  Quality of Life as measured by PROMIS Global Health Questionnaire. Total Physical Health Score of 7 to 17 with lower numbers indicating better physical health outcome and Total Mental Health Score of 8 to 16 with lower numbers indicating better mental health outcome.
Changes in Quality of Life (PROMIS Global Health Survey) | Fellowship completion [approximately 52 weeks] to 6 months post completion [approximately 77 weeks]
  Quality of Life as measured by PROMIS Global Health Questionnaire. Total Physical Health Score of 7 to 17 with lower numbers indicating better physical health outcome and Total Mental Health Score of 8 to 16 with lower numbers indicating better mental health outcome.
Changes in Self Reported Leadership Skills | Baseline to fellowship completion [approximately 52 weeks]
  The Leadership Skills Survey is designed to measure leadership skills. The survey includes 18 questions in three board types of leadership skills; administrative, interpersonal and conceptual skills. Scores will range from 6 to 30 with higher scores indicating a higher level of leaderships skills and a lower score indicating areas of leadership weakness.
Changes in Self Reported Leadership skills | Fellowship completion [approximately 52 weeks] to 6 months post fellowship completion [approximately 77 weeks]
  The Leadership Skills Survey is designed to measure leadership skills. The survey includes 18 questions in three board types of leadership skills; administrative, interpersonal and conceptual skills. Scores will range from 6 to 30 with higher scores indicating a higher level of leaderships skills and a lower score indicating areas of leadership weakness.
Changes in Burnout and Job Satisfaction | Baseline to six month post fellowship completion [approximately 77 weeks]
  The Mini Z Burnout survey is comprised of 10 items and on open ended questions. The 10 items assess satisfaction, stress, burnout, work control, chaos, values alignment, teamwork, documentation time pressure, excess electronic medical record (EMR) use at home, and EMR proficiency.
  This survey uses a 5-point likert-type scale ranging from strongly disagree (1) to strongly agree (5). Scoring for questions 1 through 10 will range from 10 to 45 with higher scores indicating a more joyful workplace and a lower score indicating burnout. The sum score for questions 1 through 4 will range from 4 to 20 with a higher score indicating a more supportive workplace and a lower score indicating a less supportive workplace. The sum of questions 5 though 8 will range from 4 to 20 with a higher score indicating an office with a good pace and manageable electronic medical record (EMR) stress and a lower score indicating a less manageable pace and more EMR stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific northwest university of health sciences, Yakima, Washington, United States